CLINICAL TRIAL: NCT06700538
Title: A Phase 1/2a Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of ARO-INHBE in Adult Volunteers With Obesity With and Without Diabetes Mellitus
Brief Title: Study of ARO-INHBE in Adults With Obesity With and Without Diabetes Mellitus
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Arrowhead Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AROINHBE-1001
Record Dates: First submitted 2024-11-20; First posted 2024-11-22 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity | interventions — Tirzepatide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (4):
- Part 1: ARO-INHBE (Experimental): ARO-INHBE in single (Day 1) or multiple (Days 1 and 29) ascending doses
  Interventions: Drug: ARO-INHBE
- Part 1: Placebo (Placebo Comparator): Placebo in single (Day 1) or multiple (Days 1 and 29) matching doses
  Interventions: Drug: Placebo
- Part 2: ARO-INHBE + Tirzepatide (Experimental): ARO-INHBE at ascending doses on Days 1 and 29 plus weekly doses of tirzepatide (2.5 to 5 mg) starting Day 15 through Day 169
  Interventions: Drug: ARO-INHBE; Drug: Tirzepatide
- Part 2: Placebo + Tirzepatide (Placebo Comparator): Placebo dose on Days 1 and 29 plus weekly doses of tirzepatide (2.5 to 5 mg) starting Day 15 through Day 169
  Interventions: Drug: Placebo; Drug: Tirzepatide

INTERVENTIONS:
Drug: ARO-INHBE — SC injection
  Arms: Part 1: ARO-INHBE; Part 2: ARO-INHBE + Tirzepatide
Drug: Placebo — calculated volume to match active treatment by SC injection
  Arms: Part 1: Placebo; Part 2: Placebo + Tirzepatide
Drug: Tirzepatide — SC injection
  Arms: Part 2: ARO-INHBE + Tirzepatide; Part 2: Placebo + Tirzepatide

SUMMARY:
This is a Phase 1/2a double-blind dose-escalating study to evaluate the safety, tolerability, pharmacokinetics (PK) and pharmacodynamics (PD) of single and multiple doses of ARO-INHBE in adult participants with obesity (Part 1), and the safety, tolerability and PD of multiple doses of ARO-INHBE in adult participants with obesity with and without type 2 diabetes mellitus receiving tirzepatide (Part 2).

ELIGIBILITY:
Inclusion Criteria:

* Obesity, defined as Body Mass Index (BMI) between 30 to 50 kg/m2 at Screening
* At least one self-reported, unsuccessful attempt at weight loss with lifestyle modification
* Willing, able and motivated to comply with all study assessments and adhere to the protocol schedule, including adherence to a stable diet and exercise routine for the duration of the study
* No abnormal finding of clinical relevance at Screening that, in the opinion of investigator, could adversely impact subject safety or adversely impact study results
* Participants of childbearing potential must agree to use highly effective contraception in addition to a condom during the study and for at least 90 days following the endo of the study or last dose of study medication, whichever is later. Participants must not donate sperm or eggs during the study and for at least 90 days following the end of the study or last dose of study medication, whichever is later.

Exclusion Criteria:

* Self-reported (or documented) weight gain or loss >5% within 3 months prior to Screening
* Use of GLP1R agonists (liraglutide, semaglutide, etc.) for any indication within 6 months prior to Screening
* Use of non-GLP1R medications for weight loss within 3 months prior to Screening, including but not limited to naltrexone/bupropion, orlistat, phentermine/topiramate, and other prescription or over-the-counter medication or supplements taken for weight loss
* Obesity attributable, in the investigator's opinion, to medication use, endocrinologic or monogenic disorders
* History or prior surgical or device-based therapy for obesity
* Use of medications strongly associated with weight gain within 3 months prior to Screening
* Type 1 diabetes mellitus
* History of hyperthyroidism or thyroid-stimulating hormone (TSH) levels <0.4 or >6.0 mIU/L at Screening
* Evidence of clinically significant end-organ disease

Note: Other Inclusion/Exclusion criteria may apply per protocol

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2024-12-04 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with Treatment-Emergent Adverse Events (TEAEs) | Part 1 single dose: up to Day 113 End of Study (EOS), Part 1 multiple doses: up to Day 169 (EOS), Part 2: up to Day 169 (EOS)

SECONDARY OUTCOMES:
Pharmacokinetics (PK) of ARO-INHBE: Maximum observed Plasma Concentration (Cmax) | Part 1: single dose (Day 1): Through 48 hours post-dose; Part 1: multiple dose (Day 1, Day 29): Through 48 hours post first and second dose
PK of ARO-INHBE: Time to Maximum Observed Plasma Concentration (Tmax) | Part 1: single dose (Day 1): Through 48 hours post-dose; Part 1: multiple dose (Day 1, Day 29)
PK of ARO-INHBE: Area Under the Plasma Concentration Versus Time Curve from Zero to 24 Hours (AUC0-24) | Part 1: single dose (Day 1): Through 48 hours post-dose; Part 1: multiple dose (Day 1, Day 29)
PK of ARO-INHBE: Area Under the Plasma Concentration Versus Time Curve from Zero to the Last Quantifiable Plasma Concentration (AUC0-t) | Part 1: single dose (Day 1): Through 48 hours post-dose; Part 1: multiple dose (Day 1, Day 29)
PK of ARO-INHBE: Area Under the Plasma Concentration Versus Time Curve from Zero to Infinity (AUC0-∞) | Part 1: single dose (Day 1): Through 48 hours post-dose; Part 1: multiple dose (Day 1, Day 29)
PK of ARO-INHBE: Terminal Half-life (t1/2) | Part 1: single dose (Day 1): Through 48 hours post-dose; Part 1: multiple dose (Day 1, Day 29)
PK of ARO-INHBE: Apparent Systemic Clearance (CL/F) | Part 1: single dose (Day 1): Through 48 hours post-dose; Part 1: multiple dose (Day 1, Day 29)
PK of ARO-INHBE: Apparent Terminal-phase Volume of Distribution (Vz/F) | Part 1: single dose (Day 1): Through 48 hours post-dose; Part 1: multiple dose (Day 1, Day 29)
PK of ARO-INHBE: Recovery of Unchanged Drug in Urine from Time 0 to 24 Hours after dosing (amount excreted: Ae) | Part 1: single dose (Day 1): Through 48 hours post-dose; Part 1: multiple dose (Day 1, Day 29)
PK of ARO-INHBE: Fraction or Percentage of Administered Drug Excreted in Urine from Time 0 to 24 Hours after Dosing (Fe) | Part 1: single dose (Day 1): Through 48 hours post-dose; Part 1: multiple dose (Day 1, Day 29)
PK of ARO-INHBE: Renal Clearance (CLr) | Part 1: single dose (Day 1): Through 48 hours post-dose; Part 1: multiple dose (Day 1, Day 29)

CONTACTS AND LOCATIONS:
Locations (3):
- New Zealand (3):
  - Research Site 1, Grafton, Auckland
  - Research Site 3, Auckland
  - Research Site 2, Christchurch

IPD SHARING:
Plan to Share IPD: No